CLINICAL TRIAL: NCT04841707
Title: Total-Body Parametric 18F-FDG PET of COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1697954
Record Dates: First submitted 2021-03-31; First posted 2021-04-12 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- COVID-19 patients (Experimental)
  Interventions: Device: uEXPLORER/mCT

INTERVENTIONS:
Device: uEXPLORER/mCT — Each participant will undergo two 18F-FDG PET/CT scans, one at baseline and one at 4- month (+/- 2 weeks) follow-up.

SUMMARY:
The primary objective is to measure the change between COVID-19 patients and normal subjects; the secondary objective is to measure the change in COVID-19 patients between baseline and 4-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive patients will have a previous positive COVID-19 test and radiographic findings, and/or a positive SARS-CoV-2 antibody test and be in early recovery.
* First PET/CT visit needs to be within 8 weeks of COVID-19 diagnosis.
* Ability to understand and willingness to sign an informed consent form.
* Ability to adhere to the study visit schedule and other protocol requirements.
* All persons ≥18 years of age.

Exclusion Criteria:

* Pregnant or lactating women.
* Any condition that would prohibit the understanding or rendering of informed consent.
* Unable to lie supine for 1-hour imaging with PET.
* Prisoners.
* Any comorbidity that, in the opinion of the investigator, could compromise protocol objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
BAB permeability assessed | 1 imaging visit up to 60 minutes
  Evaluating if there is a change in BAB permeability assessed by lung FDG K1 for patients with COVID 19

SECONDARY OUTCOMES:
4 month follow-up PET/CT scan | 1 imaging visit up to 60 minutes
  Evaluate the change in the scans between baseline scan and 4-month follow-up scan by assessing the pulmonary blood-air barrier permeability to glucose

CONTACTS AND LOCATIONS:
Overall Officials: Guobao Wang, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/total-body-parametric-18f-fdg-pet-of-covid-19-612590/

DOCUMENTS (2):
  • Study Protocol (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT04841707/Prot_000.pdf
  • Informed Consent Form (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT04841707/ICF_001.pdf